CLINICAL TRIAL: NCT05793424
Title: Establishment of a CSF Bank for the Development of Biomarkers of Smooth Muscle Cell Damage in Monogenic Cerebral Small Vessel Disease CSF-cSVD-biobank -- Constitution d'Une Banque de LCR Pour le développement de Biomarqueurs d'Atteinte Des Cellules Musculaires Lisses Dans Les Pathologies Micro-vasculaires cérébrales monogéniques CSF-cSVD-biobank
Brief Title: Establishment of a CSF Bank for the Development of Biomarkers of Smooth Muscle Cell (SMC) Damage in Monogenic Cerebral Small Vessel Disease
Acronym: CSF-cSVD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220744
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Small Vessel Diseases; CADASIL (Diagnosis)
MeSH Terms: conditions — Cerebral Small Vessel Diseases; CADASIL; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cerebral small vessel disease ( cSVD)
  Interventions: Other: Cerebrospinal fluid (CSF) sample and additional blood samples
- Control patients

INTERVENTIONS:
Other: Cerebrospinal fluid (CSF) sample and additional blood samples — Lumbar puncture (Spinal Tap) and additional blood samples
  Groups: Patients with cerebral small vessel disease ( cSVD)

SUMMARY:
The main objective of this research is to obtain biological markers of smooth muscle cells dysfunction or degeneration in cerebral small vessel diseases.

The aim of this research is therefore to build up a biocollection of CSF and blood samples from 1) patients with CADASIL disease (the most common form of cSVD) responsible for an accumulation of the NOTCH3 protein in the microvessel wall, 2) patients with other forms of monogenic cSVD (rarer) which are not responsible for an accumulation of this protein despite the damage to the smooth muscle cells of the vessel wall and 3) control patients without cSVD, collected in the context of care.

This bio-collection will allow the identification and assay of markers testifying to the damage of the smooth muscle cells (SMC) in different types of cSVD of hereditary origin, the first of which will be the soluble NOTCH3 protein.

ELIGIBILITY:
For patients woth monogenic cSVD :

Inclusion Criteria:

* Patients aged between 18 and 80 years at the time of inclusion
* Diagnosis confirmed by detection of a pathogenic mutation in the NOTCH3 gene characteristic of CADASIL, or in another gene responsible for other forms of monogenic cSVD (such as COL4A1, COL4A2, HTRA1).
* Beneficiary of a social security system
* Having given their written consent

Non inclusion Criteria:

* Contraindication to lumbar puncture:
* Haemostasis disorder (severe thrombocytopenia <60,000/mm3, PT abnormalities, INR>1.5 and/or aPTT>1.5) or anticoagulant use.
* Spinal plaque in or near the lumbar region (surgery) that may interfere with CSF collection
* Behavioural disorder that may interfere with the sampling process
* Intracranial process, intracranial hypertension or risk of involvement on imaging
* Skin lesions (inflammation or infection of any kind) or developmental abnormality (myelomeningocele) adjacent to the puncture site
* Person referred to in articles L. 1121-5 to L. 1121-8 and L. 1122-12 of the public health code, defined as :
* Pregnant, parturient or breastfeeding woman
* Person deprived of liberty by judicial or administrative decision
* Person hospitalised without consent and not subject to a legal protection measure, and person admitted to a health or social establishment for purposes other than research
* Minor
* Person of full age subject to a legal protection measure (guardianship, curators or safeguard of justice), person of full age unable to express their consent and not subject to a protection measure
* Person subject to an exclusion period for another research
* Patients participating in other interventional research
* Contraindication to lumbar puncture:
* Haemostasis disorder (severe thrombocytopenia <60,000/mm3, PT abnormalities, INR>1.5 and/or aPTT>1.5) or anticoagulant use.
* Spinal plaque in or near the lumbar region (surgery) that may interfere with CSF collection
* Spinal plaque (surgery)
* Behavioural disorder that may interfere with the sampling process
* Intracranial process, intracranial hypertension or risk of involvement on imaging
* Skin lesions (psoriasis, infection....)inflammation or infection of any kind) or developmental abnormality (myelomeningocele) adjacent to the puncture site
* Person referred to in articles L. 1121-5 to L. 1121-8 and L. 1122-12 of the public health code, defined as
* Pregnant, parturient or breastfeeding woman
* Person deprived of liberty by judicial or administrative decision
* Person hospitalised without consent and not subject to a legal protection measure, and person admitted to a health or social establishment for purposes other than research
* Minor
* Person of full age subject to a legal protection measure (guardianship, curators or safeguard of justice), person of full age unable to express their consent and not subject to a protection measure
* Person subject to an exclusion period for another research
* Patients participating in other interventional research

For control patients ( selection after CSF sampling):

Inclusion criteria :

* Subject aged 18-80 years at the time of inclusion
* Imaging done: strictly normal CT scan OR MRI showing no abnormality suggestive of cSVD
* Beneficiary of a social security system
* Having had CSF and blood samples taken as part of the treatment
* Agreement to use blood and CSF samples remainders for research purposes (information and non-opposition).
* Women who were pregnant at the time the samples were taken will not be offered to participate in the study

Non inclusion criteria :

* Any previously identified intracranial vascular pathology requiring specific management (vasculitis, acute reversible angiopathy, severe intracranial atheroma)
* Acute or chronic infectious disease (meningitis or meningoencephalitis)
* Known pregnancy
* Persons participating in other interventional research
* Preparation and freezing time for blood and CSF samples is more than 4 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients : Patients with cerebral small vessel disease (cSVD) Controls : Patients hospitalized in neurology without any cSVD
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Differential CSF proteins | At inclusion
  Differential ELISA determination of CSF proteins between monogenic cSVD patients and controls

SECONDARY OUTCOMES:
Differential blood proteins | At inclusion
  Differential ELISA determination of blood (plasma) proteins between monogenic cSVD patients and controls
Correlation blood and CSF | At inclusion
  Spearman correlation between plasma and CSF proteins assays in patients
Number | At inclusion
  Number of CSF and blood samples obtained in monogenic cSVD patients and the control population
Effect of age on blood | At inclusion
  Effect of age on ELISA determination of blood (plasma) proteins in patients and controls
Effect of age on CSF | At inclusion
  Effect of age on ELISA determination of CSF proteins in patients and controls
Link between blood protein assays and strokes | At inclusion
  Correlation between plasma proteins assays in patients on the number of strokes in patients
Link between CSF protein assays and strokes | At inclusion
  Correlation between CSF proteins assays in patients on the number of strokes in patients
Link between blood protein assays and Rankin | At inclusion
  Correlation between plasma proteins assays in patients on the modified Rankin score
  Wilson JL, Hareendran A, Hendry A, et al. (2005). "Reliability of the Modified Rankin Scale Across Multiple Raters: Benefits of a Structured Interview". Stroke. 36 (4): 777-781.
  Modified Rankin Scale permits to evaluate the degree of disability or dependance in daily activities of people who have suffered a stroke or other causes of neurological disability. It is a 6-level scale ranging from 1 to 6. The higher the score the higher the disability.
Link between CSF protein assays and Rankin | At inclusion
  Correlation between CSF proteins assays in patients on the modified Rankin score
  Wilson JL, Hareendran A, Hendry A, et al. (2005). "Reliability of the Modified Rankin Scale Across Multiple Raters: Benefits of a Structured Interview". Stroke. 36 (4): 777-781.
  Modified Rankin Scale permits to evaluate the degree of disability or dependance in daily activities of people who have suffered a stroke or other causes of neurological disability. It is a 6-level scale ranging from 1 to 6. The higher the score the higher the disability.
Link between blood protein assays and MMSE | At inclusion
  Correlation between plasma proteins assays in patients on the Mini-Mental State Examination (MMSE)
  Folstein MF, Folstein SE, McHugh PR, " Mini-mental state : a practical method for grading the cognitive state of patients for the clinician " J Psychiatr Res, 1975;12:189-198
  The Mini-Mental State Examination (MMSE) permits to evaluate cognitive state of patients. It is a 30 items scale and the score varies between 0 and 30. The higher the score the better cognitive function.
Link between CSF protein assays and MMSE | At inclusion
  Correlation between CSF proteins assays in patients on the Mini-Mental State Examination (MMSE)
  Folstein MF, Folstein SE, McHugh PR, " Mini-mental state : a practical method for grading the cognitive state of patients for the clinician " J Psychiatr Res, 1975;12:189-198
  The Mini-Mental State Examination (MMSE) permits to evaluate cognitive state of patients. It is a 30 items scale and the score varies between 0 and 30. The higher the score the better cognitive function.

IPD SHARING:
Plan to Share IPD: Undecided